CLINICAL TRIAL: NCT01009294
Title: A Phase 2a Study of Ataluren (PTC124) in Nonambulatory Patients With Nonsense-Mutation-Mediated Duchenne/Becker Muscular Dystrophy
Brief Title: Study of Ataluren (PTC124) in Nonambulatory Participants With Nonsense-Mutation-Mediated Duchenne/Becker Muscular Dystrophy (nmDMD/BMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early because a similar study with Ataluren exhibited lack of efficacy at the high dose (not due to safety concerns).
Sponsor: PTC Therapeutics (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-008-DMD; 2009-013169-24 (EudraCT Number)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Becker muscular dystrophy; Nonsense mutation; Premature stop codon; DMD; BMD; Ataluren; PTC124
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ataluren (Experimental): Ataluren was provided as a vanilla-flavored powder to be mixed with water, apple juice, or milk. Study drug dosing was based on milligrams of drug per kilogram of body weight. The dose level for ataluren was 20 milligrams/kilograms (mg/kg) in the morning, 20 mg/kg at midday, and 40 mg/kg in the evening. Administration within 30 minutes after a meal was recommended. Study drug was taken for up to 50 days.
  Interventions: Drug: Ataluren; Drug: Chronic Corticosteroid Therapy

INTERVENTIONS:
Drug: Ataluren — Oral powder
  Other Names: PTC124
Drug: Chronic Corticosteroid Therapy — Enrollment was stratified to ensure evaluation of approximately half of the participants were receiving chronic corticosteroid therapy and approximately half of participants were not receiving chronic corticosteroid therapy. Therefore, 3 out of 6 participants were receiving chronic corticosteriod therapy. For the participants receiving chronic corticosteriod therapy, a stable corticosteriod regimen was to be maintained during the study.

SUMMARY:
Duchenne/Becker muscular dystrophy (DMD/BMD) is a genetic disorder that develops in boys. It is caused by a mutation in the gene for dystrophin, a protein that is important for maintaining normal muscle structure and function. Loss of dystrophin causes muscle fragility that leads to weakness and loss of walking ability during childhood and teenage years. A specific type of mutation, called a nonsense (premature stop codon) mutation is the cause of DMD/BMD in approximately 10-15% of boys with the disease. Ataluren (PTC124) is an orally delivered, investigational drug that has the potential to overcome the effects of the nonsense mutation. This study is a Phase 2a trial that enrolled boys with nonsense mutation DMD/BMD who have lost independent mobility due to the disease. This study evaluated the safety and tolerability of ataluren (PTC124) and also evaluated efficacy outcomes in this participant population.

DETAILED DESCRIPTION:
It was planned that this Phase 2a, open-label, safety and efficacy study to be performed at 5 sites in the US and 1 site in the United Kingdom.

The study was to enroll ~30 boys with nonsense mutation DMD/BMD (nmDBMD) who have been nonambulatory for at least 1 year. Enrollment was to be stratified to ensure evaluation of ~15 participants who were receiving chronic corticosteroid therapy and of ~15 participants who were not receiving chronic corticosteroid therapy. Participants were to take ataluren 3 times per day (at breakfast, lunch, and dinner) for 48 weeks (~1 year). Study assessments were to be performed at clinic visits during screening, every 6 weeks for 2 visits and then every 12 weeks until the end of the study. Additional safety laboratory testing was to be required 4 times during the course of the study; this could have been performed at the investigational site, at an accredited local laboratory or clinic, or in the participant's home using a nursing service. When the blind for a similar study (PTC124-GD-007-DMD; NCT00592553) was revealed, the results indicated lack of efficacy for the high dose. Therefore, even though an independent data monitoring committee (DMC) agreed that both ataluren dose levels were well tolerated by the participants, the DMC recommended discontinuing ongoing studies with participants with nmDBMD receiving high-dose ataluren.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD or BMD
* Presence of a nonsense mutation in the dystrophin gene
* Unable to ambulate independently for ≥1 year due to DMD/BMD
* Presence of sufficient shoulder and elbow function to perform study-related functional procedures (for example, 9-hole peg test)
* Adequate hepatic, renal, and adrenal function
* Ability to provide evaluable pretreatment echocardiogram and lung function assessments
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions
* Ability to provide written informed consent (parental/guardian consent if applicable)/assent (if <18 years of age)

Exclusion Criteria:

* Initiation of systemic corticosteroid therapy within 6 months prior to start of study treatment or use of systemic aminoglycoside antibiotic within 3 months prior to start of study treatment
* Use of any intermittent systemic corticosteroid therapy regimen (for example, 10 days on followed by 10 days off, weekend dosing, every-other-day dosing); note that participants must have either been receiving a daily dosing regimen of prednisone, prednisolone, or deflazacort at the time of enrollment into the study or must have not been receiving any systemic corticosteroids
* Any change in treatment for congestive heart failure within 3 months prior to start of study treatment
* Ongoing warfarin or phenytoin therapy
* Prior therapy with ataluren
* Known hypersensitivity to any of the ingredients or excipients of ataluren (Litesse® UltraTM [refined polydextrose], polyethylene glycol 3350, Lutrol® micro F127 [poloxamer 407], mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, Cab O Sil® M5P [colloidal silica], magnesium stearate).
* Exposure to another investigational drug within 2 months prior to start of study treatment
* History of major surgical procedure within 1 month prior to start of study treatment or expectation of major surgical procedure (for example, scoliosis surgery) during the 48-week treatment period of the study
* Ongoing immunosuppressive therapy (other than corticosteroids)
* Ongoing participation in any other clinical trial
* Requirement for daytime ventilator assistance
* Uncontrolled clinical symptoms and signs of congestive heart failure
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings, electrocardiogram (ECG) findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow up would be completed, or could impair the assessment of study results

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male participants only are being studied.
Enrollment: 6 (Actual)
Dates: Start 2010-01-13 (Actual); Primary Completion 2010-03-23 (Actual); Study Completion 2010-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leone Atkinson, MD, PhD, Study Director — PTC Therapeutics
Locations (6):
- United States (5):
  - University of California-Davis, Davis, California
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
- University of Newcastle, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 participants with nonsense mutation Duchenne/Becker muscular dystrophy (nmDBMD) and were nonambulatory signed the informed consent form and were screened for eligibility. Six of these participants were enrolled at 2 sites. Three of the participants were receiving chronic corticosteroid therapy.
Pre-assignment Details: When the Sponsor terminated the study, the participants were told to discontinue ataluren treatment, and to return all unused ataluren to the site for return to the Sponsor. Because of difficulty of traveling to the clinic for these nonambulatory participants, the planned final visits were not performed.
Period: Overall Study
Arm/Group | Ataluren
Started | 6
Received at Least 1 Dose of Study Drug | 6
Completed | 0
Not Completed | 6
Not completed — Study discontinued by Sponsor | 6

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Ataluren: Ataluren was provided as a vanilla-flavored powder to be mixed with water, apple juice, or milk. Study drug dosing was based on milligrams of drug per kilogram of body weight. The dose level for ataluren was 20 mg/kg in the morning, 20 mg/kg at midday, and 40 mg/kg in the evening. Administration within 30 minutes after a meal was recommended. Study drug was taken for up to 50 days.
Arm/Group | Ataluren
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants]
  12 to 17 years | 3
  18 to 20 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is any untoward medical occurrence or undesirable event(s) experienced in a participant that begins or worsens following administration of the study drug or study treatment, whether or not considered related to the treatment by the Investigator. A serious adverse event (SAE) was an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason, death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), or persistent or significant disability/incapacity not related to nmDBMD. AEs included both SAEs and non-serious AEs. AEs were classified according to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE) and coded using the Medical Dictionary for Regulatory Activities (MedDRA). A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 50
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 6
Participants
  TEAEs | 1
  Treatment Emergent SAEs | 0
  AEs Related to Study Treatment | 0

2. Secondary Outcome: Time to Complete Upper Limb Function Tasks as Measured by the Jebsen Test
Description: Arm and hand function were assessed using the Jebsen test, a standardized clinical evaluation of tasks important to daily living. The test comprises of unilateral subtests performed with each hand (the dominant [DOM] hand and the non-DOM hand): moving and stacking light (250 grams) and heavy (500 grams) objects; picking up small, commonly encountered objects; stacking checkers; simulated feeding; simulated page turning; and writing. Participant performance of each task was timed. Longer time to complete the test indicates worse hand function.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable upper limb function tasks data.
Measure: Median (Full Range); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 6
seconds
  Lifting Large Heavy Objects, DOM Hand, Baseline | 11 [5 to 120]
  Lifting Large Heavy Objects, DOM Hand, Week 6: number analyzed (Participants) | 2
  Lifting Large Heavy Objects, DOM Hand, Week 6 | 10 [9 to 11]
  Lifting Large Heavy Objects, Non-DOM Hand Baseline | 11 [5 to 120]
  Lifting Large Heavy Objects, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Lifting Large Heavy Objects, Non-DOM Hand, Week 6 | 11 [7 to 14]
  Lifting Large Light Objects, DOM Hand, Baseline | 9 [4 to 120]
  Lifting Large Light Objects, DOM Hand, Week 6: number analyzed (Participants) | 2
  Lifting Large Light Objects, DOM Hand, Week 6 | 15 [7 to 22]
  Lifting Large Light Objects, Non-DOM Hand Baseline | 7 [3 to 120]
  Lifting Large Light Objects, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Lifting Large Light Objects, Non-DOM Hand, Week 6 | 12 [6 to 18]
  Stacking Large Heavy Objects, DOM Hand, Baseline | 118 [10 to 120]
  Stacking Large Heavy Objects, DOM Hand, Week 6: number analyzed (Participants) | 2
  Stacking Large Heavy Objects, DOM Hand, Week 6 | 45 [27 to 63]
  Stacking Large Heavy Objects Non-DOM Hand Baseline | 120 [28 to 120]
  Stacking Large Heavy Objects, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Stacking Large Heavy Objects, Non-DOM Hand, Week 6 | 92 [63 to 120]
  Stacking Large Light Objects, DOM Hand, Baseline | 69 [5 to 120]
  Stacking Large Light Objects, DOM Hand, Week 6: number analyzed (Participants) | 2
  Stacking Large Light Objects, DOM Hand, Week 6 | 32 [22 to 42]
  Stacking Large Light Objects Non-DOM Hand Baseline | 23 [8 to 120]
  Stacking Large Light Objects, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Stacking Large Light Objects, Non-DOM Hand, Week 6 | 69 [18 to 120]
  Lifting Small Common Objects, DOM Hand, Baseline | 16 [7 to 120]
  Lifting Small Common Objects, DOM Hand, Week 6: number analyzed (Participants) | 2
  Lifting Small Common Objects, DOM Hand, Week 6 | 19 [18 to 19]
  Lifting Small Common Objects Non-DOM Hand Baseline | 13 [8 to 120]
  Lifting Small Common Objects, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Lifting Small Common Objects, Non-DOM Hand, Week 6 | 15 [12 to 17]
  Stacking Checkers, DOM Hand, Baseline | 7 [4 to 11]
  Stacking Checkers, DOM Hand, Week 6: number analyzed (Participants) | 2
  Stacking Checkers, DOM Hand, Week 6 | 7 [6 to 7]
  Simulated Feeding, DOM Hand, Baseline | 22 [9 to 120]
  Simulated Feeding, DOM Hand, Week 6: number analyzed (Participants) | 2
  Simulated Feeding, DOM Hand, Week 6 | 40 [15 to 64]
  Simulated Feeding, Non-DOM Hand, Baseline | 38 [12 to 120]
  Simulated Feeding, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Simulated Feeding, Non-DOM Hand, Week 6 | 34 [20 to 47]
  Simulated Page Turning, DOM Hand, Baseline | 12 [4 to 24]
  Simulated Page Turning, DOM Hand, Week 6: number analyzed (Participants) | 2
  Simulated Page Turning, DOM Hand, Week 6 | 15 [9 to 21]
  Simulated Page Turning, Non-DOM Hand, Baseline | 13 [4 to 51]
  Simulated Page Turning, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Simulated Page Turning, Non-DOM Hand, Week 6 | 12 [6 to 18]
  Writing, DOM Hand, Baseline | 22 [11 to 120]
  Writing, DOM Hand, Week 6: number analyzed (Participants) | 2
  Writing, DOM Hand, Week 6 | 66 [11 to 120]
  Writing, Non-DOM Hand, Baseline | 47 [25 to 120]
  Writing, Non-DOM Hand, Week 6: number analyzed (Participants) | 2
  Writing, Non-DOM Hand, Week 6 | 78 [36 to 120]

3. Secondary Outcome: Upper Limb Function as Measured by the Brooke Upper Extremity Functional Rating Scale
Description: Upper extremity function was assessed using the Brooke Upper Extremity Functional Rating Scale, following standardized procedures. The Brooke Upper Extremity Functional Rating Scale graded arm and shoulder function from 1 to 6, with higher values indicating less function. A rating of "1" was used when the participant was able to abduct his arms in a full circle until they touch above his head, whereas a rating of "6" was used when the participant was unable to raise his hands to his mouth and had no useful function of hands.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable upper limb function tasks data.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 6
score on a scale
  Baseline | 3 [2 to 5]
  Week 6: number analyzed (Participants) | 2
  Week 6 | 3 [3 to 3]

4. Secondary Outcome: Participant Activities of Daily Living as Assessed Using the Egen Klassifikation (EK) Scale
Description: Activities of daily living after loss of ambulation were measured using the EK scale. The EK scale is an ordinal scale ranging from 0 to 30 points where 0 represents the highest level of independent function and 30 the lowest. The scale consists of 10 categories (each scored 0 to 3), involving different functional domains including 1) ability to use wheelchair, 2) ability to transfer from wheelchair, 3) ability to stand, 4) ability to balance in the wheelchair, 5) ability to move arms, 6) ability to use hands and arms when eating, 7) ability to turn in bed, 8) ability to cough, 9) ability to speak, and 10) physical well-being. The administration of the EK scale consisted of an interview of the participant to capture how he performs the tasks of daily life (as described by Categories 1 to 9) and how he perceives his wellbeing (as described by Category 10). The interviewer observed the participant and assigned the final score for the tasks that could be observed in the clinic.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable EK Scale data.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 6
score on a scale
  Ability to Use Wheelchair, Baseline | 2 [2 to 3]
  Ability to Use Wheelchair, Week 6: number analyzed (Participants) | 2
  Ability to Use Wheelchair, Week 6 | 1 [0 to 2]
  Ability to Transfer From Wheelchair, Baseline | 2 [2 to 3]
  Ability to Transfer From Wheelchair, Week 6: number analyzed (Participants) | 2
  Ability to Transfer From Wheelchair, Week 6 | 2 [2 to 2]
  Ability to Stand, Baseline | 3 [1 to 3]
  Ability to Stand, Week 6: number analyzed (Participants) | 2
  Ability to Stand, Week 6 | 2 [1 to 3]
  Ability to Balance in the Wheelchair, Baseline | 0 [0 to 3]
  Ability to Balance in the Wheelchair, Week 6: number analyzed (Participants) | 2
  Ability to Balance in the Wheelchair, Week 6 | 0 [0 to 0]
  Ability to Move Arms, Baseline | 2 [0 to 3]
  Ability to Move Arms, Week 6: number analyzed (Participants) | 2
  Ability to Move Arms, Week 6 | 1 [1 to 1]
  Ability to Use Hands/Arms When Eating, Baseline | 2 [1 to 3]
  Ability to Use Hands/Arms When Eating, Week 6: number analyzed (Participants) | 2
  Ability to Use Hands/Arms When Eating, Week 6 | 2 [1 to 2]
  Ability to Turn in Bed, Baseline | 1 [0 to 3]
  Ability to Turn in Bed, Week 6: number analyzed (Participants) | 2
  Ability to Turn in Bed, Week 6 | 1 [0 to 1]
  Ability to Cough, Baseline | 0 [0 to 0]
  Ability to Cough, Week 6: number analyzed (Participants) | 2
  Ability to Cough, Week 6 | 0 [0 to 0]
  Ability to Speak, Baseline | 0 [0 to 0]
  Ability to Speak, Week 6: number analyzed (Participants) | 2
  Ability to Speak, Week 6 | 0 [0 to 0]
  Physical Well-Being, Baseline | 0 [0 to 0]
  Physical Well-Being, Week 6: number analyzed (Participants) | 2
  Physical Well-Being, Week 6 | 1 [0 to 1]

5. Secondary Outcome: Shoulder, Elbow, and Wrist Passive and Active Range of Motion as Measured by Goniometry
Description: Goniometry was performed to test active and passive range-of motion (RoM) of the left (L) and right (R) shoulder, elbow, and wrist following standardized procedures. The observed angle for passive and active motion for each joint was measured in degrees. Greater degree of motion indicates better response.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable range of motion data.
Measure: Median (Full Range); unit: degrees
Arm/Group | Ataluren
Number analyzed (Participants) | 6
degrees
  L Elbow Extension, Supine Passive RoM, Baseline: number analyzed (Participants) | 2
  L Elbow Extension, Supine Passive RoM, Baseline | -10 [-20 to 0]
  L Elbow Extension, Supine Passive RoM, Week 6: number analyzed (Participants) | 1
  L Elbow Extension, Supine Passive RoM, Week 6 | -15 [-15 to -15]
  R Elbow Extension, Supine Passive RoM. Baseline: number analyzed (Participants) | 2
  R Elbow Extension, Supine Passive RoM. Baseline | -13 [-25 to 0]
  R Elbow Extension, Supine Passive RoM, Week 6: number analyzed (Participants) | 1
  R Elbow Extension, Supine Passive RoM, Week 6 | -20 [-20 to -20]
  L Elbow Flexion, Sitting Active RoM, Baseline | 115 [0 to 140]
  L Elbow Flexion, Sitting Active RoM, Week 6: number analyzed (Participants) | 2
  L Elbow Flexion, Sitting Active RoM, Week 6 | -10 [-20 to 0]
  R Elbow Flexion, Sitting Active RoM, Baseline | 120 [0 to 140]
  R Elbow Flexion, Sitting Active RoM, Week 6: number analyzed (Participants) | 2
  R Elbow Flexion, Sitting Active RoM, Week 6 | 70 [0 to 140]
  L Elbow Flexion, Supine Passive RoM, Baseline | 133 [120 to 140]
  L Elbow Flexion, Supine Passive RoM, Week 6: number analyzed (Participants) | 2
  L Elbow Flexion, Supine Passive RoM, Week 6 | 138 [130 to 145]
  R Elbow Flexion, Supine Passive RoM, Baseline | 135 [110 to 140]
  R Elbow Flexion, Supine Passive RoM, Week 6: number analyzed (Participants) | 2
  R Elbow Flexion, Supine Passive RoM, Week 6 | 135 [125 to 145]
  L Shoulder Abduction, Sitting Active RoM, Baseline | 18 [0 to 55]
  L Shoulder Abduction, Sitting Active RoM, Week 6: number analyzed (Participants) | 2
  L Shoulder Abduction, Sitting Active RoM, Week 6 | 0 [0 to 0]
  R Shoulder Abduction, Sitting Active RoM, Baseline | 20 [0 to 70]
  R Shoulder Abduction, Sitting Active RoM, Week 6 | 5 [0 to 10]
  L Shoulder Abduction, Supine Passive RoM, Baseline | 170 [105 to 180]
  L Shoulder Abduction, Supine Passive RoM, Week 6: number analyzed (Participants) | 2
  L Shoulder Abduction, Supine Passive RoM, Week 6 | 175 [170 to 180]
  R Shoulder Abduction, Supine Passive RoM, Baseline | 180 [120 to 180]
  R Shoulder Abduction, Supine Passive RoM, Week 6: number analyzed (Participants) | 2
  R Shoulder Abduction, Supine Passive RoM, Week 6 | 175 [170 to 180]
  L Shoulder Flexion, Sitting Active RoM, Baseline | 10 [0 to 45]
  L Shoulder Flexion, Sitting Active RoM, Week 6: number analyzed (Participants) | 2
  L Shoulder Flexion, Sitting Active RoM, Week 6 | 10 [0 to 20]
  R Shoulder Flexion, Sitting Active RoM, Baseline | 10 [0 to 80]
  R Shoulder Flexion, Sitting Active RoM, Week 6: number analyzed (Participants) | 2
  R Shoulder Flexion, Sitting Active RoM, Week 6 | 0 [0 to 0]
  L Shoulder Flexion, Supine Passive RoM, Baseline | 165 [160 to 180]
  L Shoulder Flexion, Supine Passive RoM, Week 6: number analyzed (Participants) | 2
  L Shoulder Flexion, Supine Passive RoM, Week 6 | 170 [160 to 180]
  R Shoulder Flexion, Supine Passive RoM, Baseline | 170 [150 to 180]
  R Shoulder Flexion, Supine Passive RoM, Week 6: number analyzed (Participants) | 2
  R Shoulder Flexion, Supine Passive RoM, Week 6 | 175 [170 to 180]
  L Wrist Extension, Sitting Active RoM, Baseline | 68 [20 to 80]
  L Wrist Extension, Sitting Active RoM, Week 6: number analyzed (Participants) | 2
  L Wrist Extension, Sitting Active RoM, Week 6 | 63 [55 to 70]
  R Wrist Extension, Sitting Active RoM, Baseline | 65 [30 to 90]
  R Wrist Extension, Sitting Active RoM, Week 6: number analyzed (Participants) | 2
  R Wrist Extension, Sitting Active RoM, Week 6 | 73 [70 to 75]
  L Wrist Extension, Sitting Passive RoM, Baseline | 73 [40 to 100]
  L Wrist Extension, Sitting Passive RoM, Week 6: number analyzed (Participants) | 2
  L Wrist Extension, Sitting Passive RoM, Week 6 | 73 [60 to 85]
  R Wrist Extension, Sitting Passive RoM, Baseline | 78 [55 to 90]
  R Wrist Extension, Sitting Passive RoM, Week 6: number analyzed (Participants) | 2
  R Wrist Extension, Sitting Passive RoM, Week 6 | 78 [70 to 85]
  L Wrist Flexion, Sitting Passive RoM, Baseline | 75 [35 to 95]
  L Wrist Flexion, Sitting Passive RoM, Week 6: number analyzed (Participants) | 2
  L Wrist Flexion, Sitting Passive RoM, Week 6 | 75 [60 to 90]
  R Wrist Flexion, Sitting Passive RoM, Baseline | 80 [35 to 90]
  R Wrist Flexion, Sitting Passive RoM, Week 6: number analyzed (Participants) | 2
  R Wrist Flexion, Sitting Passive RoM, Week 6 | 68 [45 to 90]

6. Secondary Outcome: Force Exerted During Elbow Flexion and Extension, Shoulder Abduction, Hand Grip, Key Grip, and Finger Pinch as Assessed by Upper Extremity Myometry
Description: Upper extremity myometry was performed using a hand-held dynamometer following standardized procedures. The measured strength (peak force) was reported in Newtons. There are 0.22 pounds (lbs) in 1 Newton and approximately 10 Newton (9.80665 Newton) in 1 kilogram (kg). The threshold/range of the hand-held dynamometer is 0 to 500 Newtons. Bilateral assessments were done, and 3 measurements were recorded from each muscle group on each side, when possible. When the measurements were done in duplicate or triplicate, the best value was used. Greater value indicates better measurement.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable upper extremity myometry data.
Measure: Median (Full Range); unit: Newton
Arm/Group | Ataluren
Number analyzed (Participants) | 6
Newton
  Left Elbow Extension, Supine, Baseline | 12 [2 to 26]
  Left Elbow Extension, Supine, Week 6: number analyzed (Participants) | 2
  Left Elbow Extension, Supine, Week 6 | 16 [14 to 18]
  Right Elbow Extension, Supine, Baseline | 12 [1 to 26]
  Right Elbow Extension, Supine, Week 6: number analyzed (Participants) | 2
  Right Elbow Extension, Supine, Week 6 | 15 [13 to 16]
  Left Elbow Flexion, Supine, Baseline | 7 [1 to 20]
  Left Elbow Flexion, Supine, Week 6: number analyzed (Participants) | 2
  Left Elbow Flexion, Supine, Week 6 | 5 [2 to 7]
  Right Elbow Flexion, Supine, Baseline | 7 [0 to 23]
  Right Elbow Flexion, Supine, Week 6: number analyzed (Participants) | 2
  Right Elbow Flexion, Supine, Week 6 | 9 [3 to 14]
  Left Finger Pinch, Sitting, Baseline | 10 [3 to 20]
  Left Finger Pinch, Sitting, Week 6: number analyzed (Participants) | 2
  Left Finger Pinch, Sitting, Week 6 | 6 [2 to 9]
  Right Finger Pinch, Sitting, Baseline | 10 [5 to 22]
  Right Finger Pinch, Sitting, Week 6: number analyzed (Participants) | 2
  Right Finger Pinch, Sitting, Week 6 | 7 [5 to 8]
  Left Hand Grip, Sitting, Baseline | 13 [5 to 23]
  Left Hand Grip, Sitting, Week 6: number analyzed (Participants) | 2
  Left Hand Grip, Sitting, Week 6 | 13 [5 to 20]
  Right Hand Grip, Sitting, Baseline | 15 [7 to 34]
  Right Hand Grip, Sitting, Week 6: number analyzed (Participants) | 2
  Right Hand Grip, Sitting, Week 6 | 23 [16 to 29]
  Left Key Grip, Sitting, Baseline | 13 [5 to 27]
  Left Key Grip, Sitting, Week 6: number analyzed (Participants) | 2
  Left Key Grip, Sitting, Week 6 | 15 [8 to 22]
  Right Key Grip, Sitting, Baseline | 11 [5 to 24]
  Right Key Grip, Sitting, Week 6: number analyzed (Participants) | 2
  Right Key Grip, Sitting, Week 6 | 18 [6 to 30]
  Left Shoulder Abduction, Sitting, Baseline | 10 [0 to 30]
  Left Shoulder Abduction, Sitting, Week 6: number analyzed (Participants) | 2
  Left Shoulder Abduction, Sitting, Week 6 | 15 [14 to 15]
  Right Shoulder Abduction, Sitting, Baseline | 12 [0 to 25]
  Right Shoulder Abduction, Sitting, Week 6: number analyzed (Participants) | 2
  Right Shoulder Abduction, Sitting, Week 6 | 14 [14 to 14]

7. Secondary Outcome: Time to Complete Hand Fine Motor Coordination and Dexterity Tasks as Measured by 9-Hole Peg Test (9HPT)
Description: Hand fine motor coordination and dexterity were assessed using the 9HPT using standardized procedures. The 9HPT is a unilateral test in which 9 pegs were placed in a board and then removed with the dominate and non-dominate hand within a 5-minute time limit. The amount of time required to put the pegs in the holes and remove them again with each hand was recorded. Each test was conducted twice per hand. Longer time to complete the test indicates worse hand fine motor coordination and dexterity.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable 9HPT data.
Measure: Median (Full Range); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 6
seconds
  Dominant Hand, Baseline | 37 [21 to 233]
  Dominant Hand, Week 6: number analyzed (Participants) | 2
  Dominant Hand, Week 6 | 38 [34 to 40]
  Non-Dominant Hand, Baseline | 40 [3 to 51]
  Non-Dominant Hand, Week 6: number analyzed (Participants) | 2
  Non-Dominant Hand, Week 6 | 37 [35 to 46]

8. Secondary Outcome: Forced Vital Capacity (FVC) as Measured by Spirometry
Description: Pulmonary function was assessed as FVC in participants by spirometry using a study-specific spirometer. Multiple tests were conducted, if needed.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable spirometry data. Data was not collected at Week 6 as no participants were evaluable at this timepoint.
Measure: Median (Full Range); unit: liters
Arm/Group | Ataluren
Number analyzed (Participants) | 6
liters
  Baseline | 1 [0.82 to 2.95]
  Week 6: number analyzed (Participants) | 0

9. Secondary Outcome: Systolic and Diastolic Function as Measured by Echocardiography With Tissue Doppler
Description: Cardiac function was assessed by echocardiography, which included standard parameters (for example, ejection fraction, left ventricle diastolic and systolic dimensions), as well as parameters integrating Doppler flow analysis with imaging to evaluate perturbations in wall motion. A standardized data collection process harmonized data from all participating institutions and allowed for centralized review.
Time Frame: Week 24 and Week 48
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable echocardiography data. Since the study was terminated early, echocardiography data were not collected after the start of study drug administration.
Arm/Group | Ataluren
Number analyzed (Participants) | 0

10. Secondary Outcome: Heart Rate as Assessed by Radial Pulse
Description: Heart rate was measured with the radial pulse. Following the Jebsen test, the participant rested for 5 minutes in a sitting position, and the heart rate for the last minute of this rest period was collected as the resting heart rate.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable heart rate data.
Measure: Median (Full Range); unit: beats per minute
Arm/Group | Ataluren
Number analyzed (Participants) | 6
beats per minute
  Baseline | 88 [72 to 120]
  Week 6: number analyzed (Participants) | 2
  Week 6 | 100 [97 to 102]

11. Secondary Outcome: Verbal Memory and Attention as Assessed by the Digit Span Task
Description: A series of digits (0-9) were presented to the participant in an auditory format only. The task had 2 parts: in the Forward Condition, the participant was requested to repeat back the digits in the order they were presented, and in the Backward Condition, he was requested to reverse the order of presentation.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable verbal memory and attention data. The test was repeated until the participant had 0 correct responses, which was up to 7 times for the Forward Condition and up to 5 times for the Backward Condition at Baseline and at Week 6.
Measure: Number; unit: correct responses
Arm/Group | Ataluren
Number analyzed (Participants) | 6
correct responses
  Forward Condition, 1 Correct Response, Baseline | 4
  Forward Condition, 1 Correct Response, Week 6: number analyzed (Participants) | 2
  Forward Condition, 1 Correct Response, Week 6 | 1
  Forward Condition, 2 Correct Responses, Baseline | 19
  Forward Condition, 2 Correct Responses, Week 6: number analyzed (Participants) | 2
  Forward Condition, 2 Correct Responses, Week 6 | 4
  Backward Condition, 1 Correct Response, Baseline | 4
  Backward Condition, 1 Correct Response, Week 6: number analyzed (Participants) | 2
  Backward Condition, 1 Correct Response, Week 6 | 2
  Backward Condition, 2 Correct Responses, Baseline | 6
  Backward Condition, 2 Correct Responses, Week 6: number analyzed (Participants) | 2
  Backward Condition, 2 Correct Responses, Week 6 | 0

12. Secondary Outcome: HRQL as Measured by the PedsQL Inventory Generic Core Scale
Description: Health-related quality of life (HRQL) was measured by the Pediatric Quality of Life Inventory (PedsQL) Inventory Generic Core Scale. The generic core module comprised of 23 questions evaluating physical, emotional, social, and school functioning. Examples of items in each of the generic core module scales included: "It is hard for me to run"; "I feel sad or blue"; "I cannot do things that other kids my age can do;" and "It is hard to pay attention in class." Each of the generic core module items was scored on a 5-point response scale from 0 (never a problem) to 4 (almost always a problem). The appropriate age-specific version was completed. PedsQL Inventory Generic Core Scale data at Week 6 is presented.
Time Frame: Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable PedsQL Inventory Generic Core Scale data at Week 6.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 2
units on a scale
  Participant-Reported, Health and Activities | 4 [0 to 4]
  Participant-Reported, Feelings | 1 [0 to 2]
  Participant-Reported, Getting along with Others | 2 [0 to 4]
  Participant-Reported, School | 1 [0 to 2]
  Parent-Reported, Physical Functioning | 4 [0 to 4]
  Parent-Reported, Emotional Functioning | 0 [0 to 2]
  Parent-Reported, Social Functioning | 1 [0 to 4]
  Parent-Reported, School Functioning | 1 [0 to 2]

13. Secondary Outcome: HRQL as Measured by the PedsQL Multidimensional Fatigue Scale
Description: HRQL was measured by the PedsQL Multidimensional Fatigue Scale. The fatigue-specific module comprised of 18 questions evaluating general fatigue, sleep/rest fatigue, and cognitive fatigue. Fatigue-specific module obtains information relating to items such as: "I feel too tired to do things that I like to do"; "I spend a lot of time in bed"; and "I have trouble remembering more than one thing at a time." Each of the fatigue-specific module items was scored on a 5-point response scale from 0 (never a problem) to 4 (almost always a problem). The appropriate age-specific version was completed. PedsQL Multidimensional Fatigue Scale data at Week 6 is presented.
Time Frame: Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable PedsQL Multidimensional Fatigue Scale data at Week 6.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 2
units on a scale
  Participant-Reported, General Fatigue | 1 [0 to 3]
  Participant-Reported, Sleep/Rest Fatigue | 1 [0 to 2]
  Participant-Reported, Cognitive Fatigue | 1 [0 to 3]
  Parent-Reported, General Fatigue | 1 [0 to 4]
  Parent-Reported, Sleep/Rest Fatigue | 0 [0 to 2]
  Parent-Reported, Cognitive Fatigue | 1 [0 to 2]

14. Secondary Outcome: HRQL as Measured by the INQoL
Description: HRQL was measured by the Individualized Neuromuscular Quality of Life Questionnaire (INQoL). The INQoL consisted of 45 questions within 10 sections. Four of the sections evaluate key muscle disease symptoms (that is, weakness, locking [myotonia], pain, and fatigue), 5 sections evaluate the degree and importance of the impact of muscle disease on particular areas of life, and 1 section asks about the positive and negative effects of treatment. A higher score indicates greater symptom impact or worse HRQL, with a range of 0-7.
Time Frame: Week 24 and Week 48
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable INQoL data. Since the study was terminated early, INQoL data were not collected.
Arm/Group | Ataluren
Number analyzed (Participants) | 0

15. Secondary Outcome: Muscle Fragility as Determined by Serum Creatine Kinase (CK) Levels
Description: Blood samples collected for chemistry assays were used to quantify serum CK concentrations. Serum CK was assessed as a potential biomarker for muscle fragility, with a reduction in serum CK considered to be a positive outcome. The reference range was based on the age of the participant.
Time Frame: Baseline and Week 6
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable CK data. Data was not collected at Week 6 for CK Levels with the reference range of 18-363 UL as no participants were evaluable at this timepoint.
Measure: Median (Full Range); unit: units/liter (U/L)
Arm/Group | Ataluren
Number analyzed (Participants) | 6
units/liter (U/L)
  CK Levels (Reference Range 18-198 U/L), Baseline: number analyzed (Participants) | 3
  CK Levels (Reference Range 18-198 U/L), Baseline | 1217 [614 to 2136]
  CK Levels (Reference Range 18-198 U/L), Week 6: number analyzed (Participants) | 1
  CK Levels (Reference Range 18-198 U/L), Week 6 | 764 [764 to 764]
  CK Levels (Reference Range 18-363 U/L), Baseline: number analyzed (Participants) | 2
  CK Levels (Reference Range 18-363 U/L), Baseline | 2605 [1413 to 3797]
  CK Levels (Reference Range 18-363 U/L), Week 6: number analyzed (Participants) | 0
  CK Levels (Reference Range 18-408 U/L), Baseline: number analyzed (Participants) | 1
  CK Levels (Reference Range 18-408 U/L), Baseline | 2343 [2343 to 2343]
  CK Levels (Reference Range 18-408 U/L), Week 6: number analyzed (Participants) | 1
  CK Levels (Reference Range 18-408 U/L), Week 6 | 2753 [2753 to 2753]

16. Secondary Outcome: Gastrocnemius Muscle Dystrophin Expression as Determined by Immunofluoresence or by Western Blotting Techniques
Description: The gastrocnemius muscle was to be biopsied from 1 leg to assess for the production of dystrophin at Week 36. The production of dystrophin was to be measured by immunofluorescene staining of the sarcolemmal membrane or by Western blotting techniques with an antibody to the C-terminal portion of the dystrophin protein (excluding revertant fibers).
Time Frame: Week 36
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable dystrophin production data. Since the study was terminated early, gastrocnemius muscle dystrophin expression data were not collected after the start of study drug administration.
Arm/Group | Ataluren
Number analyzed (Participants) | 0

17. Secondary Outcome: Study Drug Compliance
Description: Study drug compliance was assessed by the participant daily diary and quantification of used and unused study drug. Compliance was assessed in terms of the amount of drug actually taken relative to the amount that should have been taken during the study.
Time Frame: Baseline to Day 50
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable study drug compliance data.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 4
Participants
  Missed 0 Doses | 1
  Missed 1 Dose | 2
  Missed 2 Doses | 0
  Missed 3 Doses | 0
  Missed 4 Doses | 1
  Missed >5 Doses | 0

18. Secondary Outcome: Pharmacokinetics: Ataluren Plasma Exposure
Description: Blood for ataluren concentrations over a 24-hour period was to be collected on Days 2 and 3 of Week 6. Analysis of the blood samples was to be conducted using a validated high performance liquid chromatography with tandem mass spectrometry (HPLC-MS/MS) method.
Time Frame: 0, 2, 3, 6, 8, 9, 12, 14, 15, and 24 hours after the morning dose
Population: All enrolled participants who received at least 1 dose of study drug and with evaluable plasma data. Since the study was terminated early, steady state data were not collected at Week 6.
Arm/Group | Ataluren
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 50
Arm/Group | Ataluren
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=6)
Diarrhoea (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Dysuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.